CLINICAL TRIAL: NCT01885676
Title: A Pilot Randomized, Double-blind, Placebo-controlled Clinical Trial to Obtain Preliminary Data on Efficacy and Safety in the Application of PRGF-Endoret by Mesotherapy, in the Treatment of Male and Female Androgenetic Alopecia of Over 6 Months Duration.
Brief Title: Plasma Rich in Growth Factors (PRGF-Endoret)in the Treatment of Androgenetic Alopecia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: As of 12/18/2017 notification of early closure of the trial due to lack of recruitment.
Sponsor: Biotechnology Institute IMASD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTI-01D-EC/12/ALO
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PRGF-Endoret (Experimental)
  Interventions: Device: PRGF-Endoret
- Saline Solution (Placebo Comparator)
  Interventions: Other: Saline Solution

INTERVENTIONS:
Device: PRGF-Endoret — PRGF-Endoret mesotherapy micro injection.
  Arms: PRGF-Endoret
Other: Saline Solution — Saline Solution mesotherapy micro injection
  Arms: Saline Solution

SUMMARY:
* Androgenetic alopecia (AGA) or common baldness is the most common cause of hair loss in both men and women and is caused by the action of androgens in genetically predisposed individuals.
* This clinical trial was designed to evaluate the efficacy and safety of using a preparation of autologous plasma rich in growth factors (PRGF-Endoret) in the treatment of androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Androgenetic alopecia according to the following scales:
* Men: Hamilton/Norwood Scale: grades II-VI
* Women: Ludwig Scale grades I-II.
* Possibility of follow-up during the study

Exclusion Criteria:

* No androgenetic alopecia
* Telogen and anagen effluvium
* Active inflammation or infection in the intervention area
* Presence of active systemic infections.
* Background of cancerous or precancerous lesions.
* Background of connective or rheumatic diseases.
* Suffering from any serious blood disorders.
* To have undergone treatments for alopecia in the previous 6 months.
* Previous hair implants
* Intake of drugs that affect hair loss.
* Be undergoing immunosuppressive therapy and/or anticoagulants.
* Known intolerance to mesotherapy.
* Taking contraceptives containing cyproterone acetate.
* Pregnancy
* In general, any limitations that would prevent the proper application of both treatments and the right monitoring of the efficacy variables.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hair density at three months (number of hairs per cm2) | 3 months post-treatment
  Hair density (number of hairs per cm2) will be measured for each treatment group

SECONDARY OUTCOMES:
Hair Width (micrometers) | Basal, 1, 2, and 3 months post-treatment
  Hair width will be measured for each treatment group
Anagen/telogen ratio | Basal, 1, 2, and 3 months post-treatment
  Hair cycle has different phases. Two of the most important are anagen (active growth phase of hair follicles) and telogen (resting phase of the hair follicle). This secondary outcome measure allows to measure the efficacy of the PRGF-Endoret treatment.
Terminal Hair Density | Before each one of the treatments and 1, 2 and 3 months post-treatment.
  Terminal hair density will be established for each one of the treatments
Vellous hair density | Basal,1, 2 and 3 months post-treatment
  Vellous hair will be measured for each treatment group

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clínica Eduardo Anitua., Vitoria-Gasteiz, Alava
  - Centro dermatológico estético, Alicante